CLINICAL TRIAL: NCT06650514
Title: A Phase 2 Pilot Study to Evaluate the Safety and the Anti-Tumour Activity of the Myc Inhibitor OMO-103 Administered Intravenously in Patients With Advanced High-Grade Osteosarcoma
Acronym: Osteomyc
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vall d'Hebron Institute of Oncology (Other)
Collaborators: Peptomyc S.L. (Industry); Osteosarcoma Institute (Unknown); Curing Kids' Cancer Foundation (Other); Dana-Farber Cancer Institute (Other); Memorial Sloan Kettering Cancer Center (Other); Oregon Health and Science University (Other); The Morgan Adams Foundation (Unknown); The Kristen Ann Carr Fund (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHIO23003; 2024-510987-22-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-14; First posted 2024-10-21 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: Osteosarcoma; Osteosarcoma in Children
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OMO-103 (Experimental): OMO-103 administered at the recommended phase 2 dose (6.5 mg/kg as a weekly intravenous infusion in 28-day cycles)
  Interventions: Drug: OMO-103

INTERVENTIONS:
Drug: OMO-103 — OMO-103 administered at the recommended phase 2 dose (6.5 mg/kg as a weekly intravenous infusion in 28-day cycles).

SUMMARY:
This is an open-label, unicentric, single-arm Phase 2 pilot study to serve as a proof-of-concept of OMO-103 safety and activity in patients with advanced high-grade osteosarcoma.

Patients will be treated at the RP2D (6.5 mg/kg as a weekly IV infusion) of OMO-103 to estimate anti-tumour activity and further characterise the safety, tolerability, PK, and PD of OMO-103 in advanced high-grade osteosarcoma patients. Ten (10) evaluable patients will be enrolled. At least 30% of patients will be <18 years old. The first three patients 12-15 years of age will undergo additional safety monitoring.

Patients will be treated until progression by RECIST v1.1 or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Age ≥12 years at time of informed consent.
3. Histologically proven, advanced high-grade osteosarcoma not suitable for local treatments with curative intent
4. Confirmed disease progression by radiological report to at least one line of standard chemotherapy containing cisplatin and anthracycline, and no more than 2 previous lines.
5. Measurable disease as per RECIST v1.1 criteria and documented by CT/MRI (Appendix 1 - RECIST Response Criteria). NOTE: Lesions to be used as measurable disease for the purpose of response assessment must either:

   1. not reside in a field that has been subjected to prior radiotherapy, or
   2. have demonstrated clear evidence of radiographic progression since the completion of prior radiotherapy and prior to study enrolment.
6. Provision of a newly obtained tumour biopsy (either from the primary tumour or from metastases) during screening and on-treatment from all patients >16 years of age. Notes:

   * The identified lesion to be biopsied should not have been previously irradiated and should not be the only lesion being used as a measurable-disease target lesion for objective response assessment. Patients must have tumour lesions that can be accessible for biopsy with acceptable clinical risk in the judgement of the Investigator.
   * In case a patient has had a tumour biopsy in the previous 6 months and a paraffin block is available, a new biopsy does not need to be done at Screening (if they have received no treatment after biopsy).
7. Documented progression on or following the last line of therapy.
8. ECOG performance status 0-2 (Appendix 2 - Performance Status Criteria).
9. Life expectancy of ≥ 12 weeks as estimated by the treating physician.
10. Resolution of all acute, reversible toxic effects of prior therapy or surgical procedure to Grade ≤1 (except alopecia and peripheral neuropathy to Grade ≤2).
11. Adequate organ function.
12. If not postmenopausal or surgically sterile, female patients and female sexual partners of male patients must be willing to use at least one highly effective method of birth control (hormonal contraception, IUD, abstinence, condom) for at least a menstrual cycle before and for 3 months after last study drug administration.

Exclusion Criteria:

1. Treatment with systemic anti-cancer therapy within three weeks prior to study drug administration for chemotherapy and 5 half-lives for targeted therapies.
2. Radiation therapy within four weeks prior to study entry. Localised palliative radiotherapy to nontarget lesions is allowed
3. Low-grade osteosarcoma, parosteal, or periosteal osteosarcoma.
4. Prior history of other malignancies other than osteosarcoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) unless the patient has been free of the disease for at least 2 years.
5. Non-malignant systemic disease including cerebrovascular accident, unstable angina pectoris, unstable atrial fibrillation, unstable cardiac arrhythmia, myocardial infarction in the last six months, New York Heart Association (NYHA) Class III or IV heart failure (Appendix 5 - New York Heart Association Criteria).
6. Patients with active uncontrolled infection or known to be serologically positive for human immunodeficiency virus (HIV), hepatitis B (except after vaccination) or hepatitis C infection. Investigators may test as per their discretion.
7. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.
8. Patients with symptomatic or unstable central nervous system primary tumour or metastases and/or sarcomatous meningitis
9. Live vaccine in the last four weeks.
10. Current participation in another interventional therapeutic trial.
11. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study.
12. Knowledge of any other disease or medication that may interfere with study treatment.
13. Patients with known allergies or hypersensitivity reactions to the active substance or to any of its excipients
14. Patient unable to comply with the study protocol owing to psychological, social (lack of social support or social exclusion) or geographical reasons.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Preliminary anti-tumour activity of OMO-103 monotherapy in patients with high-grade osteosarcoma | 16 weeks from start of treatment
  Progression-free survival rate at 16 weeks (16-week PFS)

SECONDARY OUTCOMES:
Further evaluate the anti-tumour activity of OMO-103 monotherapy in patients with high-grade osteosarcoma. | Until disease progression, unacceptable toxicity, patient request, physician's decision to withdraw treatment, subsequent anticancer therapy, or death whichever occurs first, assessed up to 24 months
  • Objective Response Rate (ORR) is defined as the percentage of patients with a complete response (CR) or a partial response (PR) by Investigator according to RECIST 1.1 in solid tumours.
Further evaluate the anti-tumour activity of OMO-103 monotherapy in patients with high-grade osteosarcoma. | Until disease progression, unacceptable toxicity, patient request, physician's decision to withdraw treatment, subsequent anticancer therapy, or death whichever occurs first, assessed up to 24 months
  • Disease Control Rate (DCR) is defined as the percentage of patients in whom the best overall response is determined as CR, PR, or stable disease (SD) by the Investigator according to RECIST 1.1 in solid tumours.
Further evaluate the anti-tumour activity of OMO-103 monotherapy in patients with high-grade osteosarcoma. | Until disease progression, unacceptable toxicity, patient request, physician's decision to withdraw treatment, subsequent anticancer therapy, or death whichever occurs first, assessed up to 24 months
  • Time to Response (TTR) is defined as the time from start of treatment to the date of first documentation of CR, or PR.
Further evaluate the anti-tumour activity of OMO-103 monotherapy in patients with high-grade osteosarcoma. | Until disease progression, unacceptable toxicity, patient request, physician's decision to withdraw treatment, subsequent anticancer therapy, or death whichever occurs first, assessed up to 24 months
  • Time to Progression (TTP) is defined as the time from start of treatment to the date of first documentation of disease progression.
Further evaluate the anti-tumour activity of OMO-103 monotherapy in patients with high-grade osteosarcoma. | Until disease progression, unacceptable toxicity, patient request, physician's decision to withdraw treatment, subsequent anticancer therapy, or death whichever occurs first, assessed up to 24 months
  • Duration of Response (DOR) refers to the minimum from the time when complete response (CR) or partial response (PR) is first observed to the time of progressed disease (PD)
Further evaluate the anti-tumour activity of OMO-103 monotherapy in patients with high-grade osteosarcoma. | Until patient request or death whichever occurs first, assessed up to 24 months
  • Overall survival (OS) is defined as the time from the date of start of treatment to the date of death due to any cause. Patients without documentation of death at the time of analysis will be censored at the date last known to be alive.
Safety and tolerability profile of OMO-103 monotherapy in patients with high-grade osteosarcoma. | Unrtil end of treatment assessed up to 24 months
  Incidence and severity of adverse events (AEs), graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.
Assess the benefit/risk ratio associated with OMO-103 | Until progression assessed up to 24 months
  Q-TWiST approach (Quality-adjusted Time Without Symptoms of disease recurrence or Toxicity of treatment)time experiencing toxicity (grade 3/4 AEs) before progression, time without toxicity or symptoms of progression, and time after progression
To characterise the pharmacokinetics (PK) of OMO-103 monotherapy in patients with high-grade osteosarcoma (12-15 years of age). | During the first cycle of treatment (4 weeks)
  PK parameters of OMO-103: AUC (Area Under the Curve)
To characterise the pharmacokinetics (PK) of OMO-103 monotherapy in patients with high-grade osteosarcoma (12-15 years of age). | During the first cycle of treatment (4 weeks)
  PK parameters of OMO-103: Cmax (Peak Plasma Concentration)
To characterise the pharmacokinetics (PK) of OMO-103 monotherapy in patients with high-grade osteosarcoma (12-15 years of age). | During the first cycle of treatment (4 weeks)
  PK parameters of OMO-103: tmax (time to peak drug concentration)
To characterise the pharmacokinetics (PK) of OMO-103 monotherapy in patients with high-grade osteosarcoma (12-15 years of age). | During the first cycle of treatment (4 weeks)
  PK parameters of OMO-103: t1/2 (elimination half life)
Evaluate quality of life (QoL) in patients with high-grade osteosarcoma | Unitl end of treatment assessed up to 24 months
  For adult patients: Health-related quality of life (HRQoL) measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 items (EORTC-C30)
Evaluate quality of life (QoL) in patients with high-grade osteosarcoma | Unitl end of treatment assessed up to 24 months
  For patients between 12 and 17 years of old Health-related quality of life (HRQoL) measured by the Pediatric Quality of Life Inventory (PedsQL)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided